CLINICAL TRIAL: NCT03130452
Title: Helicobacter Pylori Eradication Rates of Concomitant Therapy and Tailored Therapy Based on 23S Ribosomal RNA Point Mutations Associated With Clarithromycin Resistance: A Multicenter Prospective Randomized Study
Brief Title: Helicobacter Pylori Eradication Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Inje University (Other)
Responsible Party: Principal Investigator, Kim Ji Hyun, Clinical Professor, Inje University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-09-0025
Record Dates: First submitted 2017-04-05; First posted 2017-04-26 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Helicobacter Pylori Infection
MeSH Terms: interventions — Lansoprazole; Amoxicillin; Amoxicillin-Potassium Clavulanate Combination; Clarithromycin; Metronidazole

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- concomitant group (Active Comparator): lansoprazole 30 mg tablet, amoxicillin 1.0 g tablet, metronidazole 500 mg tablet and clarithromycin 500 mg tablet by mouth every 12 hours for 2 weeks, regardless of 23S ribosomal RNA point mutation.
  Interventions: Drug: Lansoprazole 30mg; Drug: Amoxicillin 1.0g Tab; Drug: Clarithromycin 500mg; Drug: Metronidazole 500 mg
- tailored treatment group I (Experimental): 23S ribosomal RNA point mutation negative, lansoprazole 30 mg, amoxicillin 1.0 g, and clarithromycin 500 mg were administered twice a day for 2 weeks.
  Interventions: Drug: Lansoprazole 30mg; Drug: Amoxicillin 1.0g Tab; Drug: Clarithromycin 500mg
- tailored treatment group II (Experimental): 23S ribosomal RNA point mutation positive, lansoprazole 30 mg, amoxicillin 1.0 g and metronidazole 500 mg For 2 weeks.
  Interventions: Drug: Lansoprazole 30mg; Drug: Clarithromycin 500mg; Drug: Metronidazole 500 mg

INTERVENTIONS:
Drug: Lansoprazole 30mg — lansoprazole 30 mg tablet
  Other Names: langton
Drug: Amoxicillin 1.0g Tab — Amoxicillin 1.0g tablet
  Other Names: amoxiclav
  Arms: concomitant group; tailored treatment group I
Drug: Clarithromycin 500mg — Clarithromycin 500mg tablet
  Other Names: clavacin
Drug: Metronidazole 500 mg — Metronidazole 500 mg tablet
  Other Names: lysinyl
  Arms: concomitant group; tailored treatment group II

SUMMARY:
The purpose of this study was to evaluate the efficacy and compliance of tailored therapy which using the polymerase chain reaction for point mutation of clarithromycin, compared to concomitant therapy, in patients without history of H. pylori eradication.

DETAILED DESCRIPTION:
Purpose of Study>

1. To evaluate the efficacy of tailored therapy compared to concomitant therapy.
2. Difference in eradication rate according to the frequency of 23S ribosomal RNA point mutation in clarithromycin.
3. To evaluate the compliance of tailored therapy compared to concomitant.
4. To analysis of factors which influence to the eradication rate.

Patients>

; Target disease

* peptic ulcers(gastric ulcer, duodenal ulcer),
* gastric MALToma,
* Endoscopic therapy state of early gastric cancer or gastric adenoma,
* Patients who require H. pylori testing by clinical judgment, such as chronic gastritis.

Method>

Patients with H. pylori infection who have been screened for a 23S ribosomal RNA point mutation (A2142G, A2143G point mutation) and randomized to a concomitant treatment group and a tailored treatment group. In concomitant treatment group, lansoprazole 30 mg, amoxicillin 1.0 g, metronidazole 500 mg and clarithromycin 500 mg were administered twice a day for 2 weeks, regardless of 23S ribosomal RNA point mutation. In tailored treatment group, In the case of 23S ribosomal RNA point mutation negative, lansoprazole 30 mg, amoxicillin 1.0 g, and clarithromycin 500 mg were administered twice a day for 2 weeks. In tailored treatment group, In point mutation positive cases, lansoprazole 30 mg, amoxicillin 1.0 g and metronidazole 500 mg For 2 weeks. For each treatment group, at least 4 weeks after completion of drug administration, confirm the sterilization and confirm the compliance and adverse effects of the drug.

ELIGIBILITY:
Inclusion Criteria:

* H. pylori infection diagnosed patient, between 18 years old and 80 years old
* No history of H. pylori eradication therapy
* No antibiotic use for more than 3 days within 1 month of treatment

Exclusion Criteria:

* History of taking antibiotics for more than 3 days in the last 1 month
* History of subtotal or partial gastrectomy
* Patients with other systemic disorders such as severe liver function, kidney function, cardiopulmonary function abnormality
* Pregnant and lactating women
* Disagree with the survey or do not respond to the questionnaire
* Contraindications for each medications

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 423 (Actual)
Dates: Start 2016-12-17 (Actual); Primary Completion 2019-01-28 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Comparison of success rate of H. pylori eradication between tailored therapy and concomitant therapy. | At 4 weeks after the completion of drug administration, the urea breath test is performed to check for eradication, Before the urea breath test, the proton pump inhibitor or H2 blocker should be discontinued for 2 weeks.
  Comparison of percentage of people who succeeded in H. pylori eradication among all participants in each treatment group (tailored therapy vs concomitant therapy)

SECONDARY OUTCOMES:
Difference in eradication rate according to the frequency of 23S ribosomal RNA point mutation in clarithromycin | Before the treatment, 23S ribosomal RNA point mutation is confirmed and at least 4 weeks after the end of treatment, urea breath test is performed to check whether or not eradication is completed.
  Identify the effect of 23S ribosomal RNA point mutation on the eradication rate regardless of the administration drug.

OTHER OUTCOMES:
Number of remaining medicines of tailored therapy compared to concomitant therapy | At 4 weeks after the completion of drug administration, when the patient visited for the urea breath test, check the number of remaining medicines.
  After taking the treatment drug, take out all remaining medicine in the outpatient clinic room, check the number of remaining medicines, and judge compliance.

CONTACTS AND LOCATIONS:
Overall Officials: Ji Hyun Kim, Principal Investigator — Inje University Busan Paik hosipital
Locations (1):
- Inje University Busan Paik hosipital, Busan, South Korea

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual patient data available to other researchers.